CLINICAL TRIAL: NCT00015990
Title: Phase II Study of Thalidomide in the Treatment of Myelodysplastic Syndromes in Adults: A Clinical and Biologic Study
Brief Title: Thalidomide in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01856; N998B; U10CA025224 (NIH); CDR0000068580 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-05-06; First posted 2004-02-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Refractory Anemia With Ringed Sideroblasts; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — Thalidomide

ARMS (1):
- Treatment (thalidomide) (Experimental): Patients receive oral thalidomide once daily. Treatment continues for 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: thalidomide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: thalidomide — Given orally
  Other Names: Kevadon; Synovir; THAL; Thalomid
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of thalidomide in treating patients who have myelodysplastic syndrome. Thalidomide may improve the immune system's ability to fight myelodysplastic syndrome

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine whether thalidomide improves cytopenias in patients with myelodysplastic syndromes.

II. Determine the toxicity of this regimen in these patients. III. Determine whether this regimen down regulates the peripheral blood levels of tumor necrosis factor alpha, interferon gamma, and interleukin-12 and whether these changes correlate with clinical response in these patients.

IV. Determine whether this regimen alters the peripheral blood T-cell subset distribution and whether these changes correlate with clinical response in these patients.

V. Determine the effect of this regimen on bone marrow microvessel density and whether these effects correlate with clinical response in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prognosis (favorable vs unfavorable). (Favorable stratum closed to accrual 12/28/01)

Patients receive oral thalidomide once daily. Treatment continues for 5 years in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for 1 year and then annually for 4 years.

PROJECTED ACCRUAL: A total of 20-58 patients (10-29 per stratum) will be accrued for this study within 20 months. (Favorable stratum closed to accrual 12/28/01)

ELIGIBILITY:
Inclusion Criteria:

* Pre-transfusion hemoglobin =< 10 g/dL
* Pre-transfusion platelet count =< 50,000/μL
* Absolute neutrophil count < 1000/μL
* Total bilirubin ≤ 1.5 x UNL
* Alkaline phosphatase ≤ 3 x UNL
* AST ≤ 3 x UNL
* Creatinine ≤ 1.5 x UNL
* A diagnosis of MDS as demonstrated in the bone marrow; any subtypes are eligible including:

  * Refractory anemia (cytopenia)
  * Refractory anemia with ringed sideroblasts
  * Chronic myelomonocytic leukemia
  * Refractory anemia with excess blasts
  * Refractory anemia with excess blasts in transformation
  * Unclassified MDS
* Patients with refractory anemia with excess blasts in transformation who are not candidates for (or who decline) induction chemotherapy are eligible; those patients who were candidates for (and accepted) induction chemotherapy should have failed at least 1 chemotherapy regimen prior to entry
* Patients who are candidates for marrow transplantation should have this option discussed prior to study entry

Exclusion Criteria:

* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential or their sexual partners who are unwilling to employ 2 adequate methods of contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
* Peripheral neuropathy (by history or clinical exam)
* Concomitant therapy ≤ 30 days for myelodysplastic syndrome with any specific agent including chemotherapy, corticosteroids and/or growth factors (i.e. erythropoietin, G-CSF, GM-CSF, thrombopoietic agent); patients on chronic low-dose corticosteriods (< 20 mg/d) for reasons other than MDS are allowed
* Uncontrolled infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2001-04; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Confirmed response defined as complete hematologic response (CHR) or partial response (PR) or hematological improvement (HI) on 2 consecutive evaluations in terms of proportion of successes measured using criteria reported by Cheson et al | Up to 3 months
  Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Incidence and severity of toxicities, graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to 5 years

SECONDARY OUTCOMES:
Survival time | Time from registration to death due to any cause, assessed up to 5 years
  Estimated using the method of Kaplan-Meier.
Time to disease progression | Time from registration to documentation of disease progression, assessed up to 5 years
  Estimated using the method of Kaplan-Meier.
Duration of response measured using criteria reported by Cheson et al | Date at which the patient's objective status is first noted to be either a CHR or PR to the date progression is documented, assessed up to 5 years
Time to treatment failure | Time from the date of registration to the date at which the patient is removed from treatment due to progression, toxicity, or refusal, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Moreno Aspitia, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States